CLINICAL TRIAL: NCT04763187
Title: Influence of PRGF and PRF on Post-extractive Alveolus Regeneration. Randomised Controlled Trial
Brief Title: Post-extractive Alveolus Regeneration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Valdonė Brazdeikytė, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LSMU123
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Chronic Periodontitis Apical; Embedded Tooth
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Lower molar extraction and filling of post-extraction alveolus with hemostatic sponge containing gentamicin.
  Interventions: Procedure: Tooth extraction
- PRGF group (Experimental): Post-extraction alveolus is filled with PRGF.
  Interventions: Procedure: Tooth extraction
- PRF group (Experimental): Post-extraction alveolus is filled with PRF.
  Interventions: Procedure: Tooth extraction

INTERVENTIONS:
Procedure: Tooth extraction — Tooth extraction and alveolus regeneration with autologous blood concentrate.

SUMMARY:
Healing of post-extraction alveolus is a complex process that involves soft and hard tissues regeneration. Pain, swelling, difficulty of opening the mouth, delayed healing of bone tissue, alveolitis and horizontal or vertical resorption of bone tissue are the main problems that have impact on consequent treatment. Blood concentrates PRGF (plasma rich in growth factors) and PRF (platelet-rich fibrin), which are rich in growth factors, create better conditions for post-extraction alveolus healing and enhance quality of soft tissues and bone regeneration. Our study objective was to compare physiological healing of post-extraction zone, PRF and PRGF induced changes of healing process. Methods that we used: 43 patients were randomly divided into 3 groups: I control group - lower molar extraction and filling of post-extraction alveolus with hemostatic sponge containing gentamicin, II group - post-extraction alveolus is filled PRGF and III group - post-extraction alveolus is filled with PRF. Bone regeneration was evaluated in CBCT scans after 1 month. Pain was evaluated using visual analogical scale (VAS).

DETAILED DESCRIPTION:
This was a prospective, single-centre, with unequal randomisation ratio [1,9:1:1], parallel, multiple-group (control and two experimental groups) study. Randomized clinical trial was conducted between September 2019 and December 2019 at department of Maxillofacial Surgery Clinic of Kaunas Clinics. Permission of Bioethics Center was acquired for this study. Participants of this study were patients who needed extraction of lower molars due to K04.5 (chronic apical periodontitis) and K01.0 (embedded teeth) diagnoses, based on ICD-10-CM classification. In this study participated 43 patients: 33 (76,7%) women and 10 (23,3%) men, average age - 28,6 years, the youngest was 18 years old and the oldest was 48 years old. All patients were introduced to the study protocol and gave informed consent. Confidentiality of subjects is assured because only summarized results will be published.

Patients were randomised into 3 groups: I control group - lower molar extraction and filling of post-extraction alveolus with hemostatic sponge containing gentamicin, II group - post-extraction alveolus is filled PRGF and III group - post-extraction alveolus is filled with PRF. Randomization sequence was created using Excel 2019 (Microsoft, Redmond, WA, USA) with a 1,9:1:1 allocation using random block sizes of 2 and 4. Surgery was performed by the same surgeon. After procedures of tooth extraction and PRGF or PRF application, zone of surgery was closed up using resorbable thread (Ethicon Coated Vicryl Plus 4-0) and applying the method of cross mattress suture. During procedure control group was administred with local antibiotics (gentamicin) to avoid infection possibility. Non-steroidal anti-inflammatory medication was administered one hour after procedure and before sleep. Threads were removed after 7 days. Pain felt on 1st and on 7th day after procedure was evaluated using visual analogical scale (hereinafter - VAS) during the same appointment. Pacients selected number from 0 to 10, there accordingly 0 - no pain, 5 - moderate pain and 10 - worst pain. [22] Cone beam computed tomography (hereinafter - CBCT) (E-WOO, Picasso Trio, Republic of Korea) was carried out immediately after procedure and 1 month after procedure for evaluation of bone tissue regeneration. It was decided to evaluate bone regeneration in CBCT scans (Ez3D Plus Professional Ver.1.2.6.1) at following dimensions: horizontal AA (X) (mm) and vertical AA (Y) (mm) dimensions of alveolar ridge were measured. Also, horizontal X (mm), vertical Y (mm) and diagonal Z (mm) dimensions of primary bone tissue formed in post-extraction alveolus in 1 month (Figure 2) All measurements carried out by the same examinator.

Sample size of this study was calculated by using Paniotto formula. During the research period (September to December 2019) was estimated that on average within 4 months 48 pacients applies to department of Maxillofacial Surgery Clinic of Kaunas Clinics due to lower molars extraction. After calculations with 95% probability and 0,05 error defined required sample size - 43 pacients.

Statistical analysis carried out using SPSS (Statistical Package for the Social Science for Windows; Chihago, USA) package 22.0. The diagnostic and demographic charasteristics were compared using Wilcoxon test, Kruskal-Wallis test, Mann-Whitney test and Spearman correlation analysis. Level of significance p was set at 0,05 for verification of statistical hypotheses.

Blood of 11 patients (3 men and 8 women, average age 27 years) taken from peripheral vein, using 21G blood collection needle and PRGF-Endoret® test tubes with volume of 9 ml, for production of PRGF. As per instruction of manufacturer, tubes contain 3,8 % sodium citrate, which serves as anticoagulant. In order to produce the PRGF, test tubes were centrifuged for 8 minutes in 580 g Endoret® (PRGF®) System V centrifuge. 3 different layers are formed - erythrocytes, leukocytes and blood plasma. Layer of blood plasma is divided into two fractions. 1st fraction is called plasma poor in growth factors, which forms a top layer in a tube down to 2nd fraction. 2nd fraction (2 ml of blood plasma, which is above the layer of leukocytes), forms the layer of plasma rich in growth factors. Activation of this fraction is carried out using sterile 10 % calcium chloride solution (50 µL of activator for 1 ml of blood plasma), which carried out degranulation of platelets and therefore released growth factors. After activation, test tubes were incubated at 37°C for 30 minutes, in order give the consistency of gelatin to PRGF. Formed fold or fluid was inserted into alveolus of extracted tooth, then the edges were closed up using resorbable cross mattress suture.

Blood of 11 patients (2 men and 9 women, average age 26 years) were collected from peripheral vein using 21G blood collection needle and PRF test tubes with volume of 9 ml, for production of PRF. Test tube was inserted into A-PRF centrifuge "A-PRF 12". The lid was closed and program at 2800 rpm for 12 minutes was initiated. A-PRF fold was separated from red blood cells (blood clots) in the test tube. After pulling the fold out of test tube, it was formed on sterile surgical tray. Formed fold was inserted into alveolus of extracted tooth and edges of wound were closed up using resorbable cross mattress suture.

ELIGIBILITY:
Inclusion Criteria:

* Patients who need lower molar extraction
* Patients who belong to working age group (18-50 years)

Exclusion Criteria:

* Pregnant women and postmenopausal women
* Children and older than 50 years old patients
* Oncological diseases, undergone chemotherapy and radiation therapy
* Chronic diseases
* Hormonal imbalances
* Somatic symptom disorder
* Osteoporosis, osteonecrosis
* Taking bisphosphonates, antidepressants, psychotropic drugs
* Smoking
* Psychologically dissabled patients

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Post operative pain | First day after surgery.
  Pain was evaluated using visual analogical scale (VAS). Pacients selected number from 0 to 10, there accordingly 0 - no pain, 5 - moderate pain and 10 - worst pain.
Post operative pain | Seventh day after surgery.
  Pain was evaluated using visual analogical scale (VAS). Pacients selected number from 0 to 10, there accordingly 0 - no pain, 5 - moderate pain and 10 - worst pain.
Bone regeneration | Immediately after surgery.
  Bone regeneration was evaluated in CBCT scans. In CBCT scans (Ez3D Plus Professional Ver.1.2.6.1) immediately after surgery horizontal (mm) and vertical (mm) dimensions of alveolar ridge were measured.
Bone regeneration | 1 month after surgery.
  Bone regeneration was evaluated in CBCT scans. In CBCT scans (Ez3D Plus Professional Ver.1.2.6.1) 1 month after surgery horizontal (mm) and vertical (mm) dimensions of alveolar ridge were measured. Also, horizontal (mm), vertical (mm) and diagonal (mm) dimensions of primary bone tissue formed in post-extraction alveolus in 1 month.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Pavel Rokicki, Study Director — Oral surgeon
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No